CLINICAL TRIAL: NCT02326779
Title: Low-dose Aspirin Therapy for Stage II-III Esophageal Cancer- A Multi-Center, Open Label, Randomized Controlled Phase III Trial
Brief Title: Low-dose Aspirin Therapy for Esophageal Cancer
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Why Stopped: The study could not be performed.
Sponsor: Zhejiang University (Other)
Responsible Party: Principal Investigator, Yihua, Wu, Instructor, Zhejiang University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NNSFC 81302455
Record Dates: First submitted 2014-12-22; First posted 2014-12-29 (Estimated); Last update posted 2021-04-27 (Actual); Status verified 2021-04

CONDITIONS: Esophageal Cancer
Keywords: esophageal cancer; aspirin; survival
MeSH Terms: conditions — Esophageal Neoplasms | interventions — Aspirin

ARMS (2):
- Experimental Arm (Experimental): Experimental Arm: acetylsalicylic acid (Aspirin) 100 mg OD for 3 years
  Interventions: Drug: Acetylsalicylic acid
- Comparator Arm (No Intervention): Non-aspirin use arm as comparator

INTERVENTIONS:
Drug: Acetylsalicylic acid — Acetylsalicylic acid (Aspirin) 100 mg OD for 3 years
  Other Names: Aspirin
  Arms: Experimental Arm

SUMMARY:
The aim of this study is to evaluate the survival benefit of low-dose aspirin use for stage II-III esophageal cancer patients.

DETAILED DESCRIPTION:
The investigators aimed to evaluate the hypothesis that low-dose aspirin can improve survival in stage II-III esophageal cancer patients, and to evaluate whether this effect is influenced by PIK3CA, KRAS, BRAF mutation and COX-2 expression. Eligible participants will be randomized to either aspirin treatment arm (100 mg aspirin OD for 3 years), or non-aspirin user arm in 1:1 ratio. After randomization, participants will receive 3 monthly assessments during treatment and follow-up.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female subjects with an age of 18 years or older.
2. Subjects with Stage II-III histological proven esophageal cancer.
3. Subjects with performance status (PS) of 0-1 or ECOG performance status 0-2.
4. Subjects must have signed an approved informed consent prior to any study procedures.
5. Subjects with adequate bone marrow, hepatic and renal functions, with a) neutrophils ≥ 1.5x109/ L; platelets ≥ 100x109/L; hemoglobin ≥ 9g/dL; b) Total bilirubin ≤ 2.0 x the upper limit normal; ALT and AST ≤ 2.5 x ULN (≤ 5 x ULN in case of liver metastasis); c) creatinine clearance > 50 ml/min;
6. Subjects undergone complete resection of primary tumor;
7. Subjects with life expectancy ≥ 3 months.
8. Completed standard therapy ( at least 3 months of chemotherapy ± radiotherapy )
9. Within 120 days of completion of standard therapy (surgery, chemotherapy ± radiotherapy)

Exclusion Criteria:

1. Subjects with haemorrhagic diathesis (i.e. haemophilia).
2. Subjects with prior malignant tumors except for esophageal cancers in the past 5 years.
3. Subjects with documented or suspected central nervous system metastases.
4. Subjects with serious, nonhealing wound, ulcer, or bone fracture.
5. Subjects with a history of stroke, coronary arterial disease, angina, or vascular disease.
6. Subjects who are pregnant, lactating, or not using adequate contraception.
7. Subjects who have known allergy to NSAID or Aspirin.
8. Subjects receiving other antiplatelet agents (i.e. clopidogrel, ticlopidine) or anticoagulants (i.e. warfarin, low molecular weight heparins).
9. Subjects receiving current long term treatment (≥ 1 month) with Aspirin or other NSAIDs.
10. Subject unwilling or unable to comply with study requirements.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2016-03; Primary Completion 2018-10 (Estimated); Study Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
Disease-free survival | 5 years
Overall survival | 5 years

SECONDARY OUTCOMES:
Adverse events | 5 years